CLINICAL TRIAL: NCT00769314
Title: A Randomised, Double-Blind, Single Dose, One-Day Early Administration, Multicentre Study Comparing the Efficacy and Safety of Acyclovir Lauriad® 50 mg Muco-adhesive Buccal Tablet to Matching Placebo, in the Treatment of Herpes Labialis in Immunocompetent Patients.
Brief Title: Phase 3 Clinical Study for the Treatment of Cold Sore
Acronym: LIP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valerio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BA2005/21/02
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Results first posted 2012-12-21 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-11

CONDITIONS: Herpes Labialis
MeSH Terms: conditions — Herpes Labialis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Acyclovir Lauriad 50mg
  Interventions: Drug: Acyclovir Lauriad
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acyclovir Lauriad — 50 mg muco-adhesive buccal tablets, single application on the gum
  Arms: 1
Drug: Placebo — 50 mg muco-adhesive buccal tablets, single application on the gum
  Arms: 2

SUMMARY:
To demonstrate the efficacy of a single dose of acyclovir Lauriad® 50mg muco-adhesive buccal tablet versus a single dose of matching placebo on the primary vesicular lesion of cold sore.

ELIGIBILITY:
Inclusion Criteria:

* History of recurrent herpes labialis lesions where:

  * At least 50% of previous episodes produced classical lesions to the vesicular stage (i.e. episodes that progressed through macula, papule, vesicle, crust and healed);
  * Prodromal symptoms (itching, tingling, pain etc.) should precede herpes labialis lesions in at least 50% of the previous herpes episodes
* Good general health (ECOG < 2), immunocompetent
* Signed and dated written informed consent
* Women of childbearing potential must have effective contraception method

Exclusion Criteria:

* More than 50% of recurrences that aborted spontaneously in the past 12 months
* Primary herpes lesion outside the lips (e.g. nose, chin, etc.)
* Abnormal peri-oral skin condition that might affect the normal course of cold sores (e.g. eczema, psoriasis…)
* Oral diseases whose prodromal symptoms may mimick those of herpes labialis, including recurrent oral aphthous disease
* Oral diseases that might interfere with the evaluation of the efficacy or safety of the treatments, including gingivitis, parondotis, mucositis, oropharyngeal candidiasis…
* History of infection known to be resistant to acyclovir family agents
* Previous vaccination against herpes
* Concomitant treatment likely to interfere with acyclovir
* Allergy to any acyclovir containing agents
* Immunocompromised condition, including HIV+
* Unability to properly understand protocol requirements, to follow the study procedures, to complete the patient diary or to start the self-initiation of the treatment
* Upper full or partial dentures with acrylic border in the canine fossa
* Milk allergy or known history of hypersensitivity to one of the components of the products
* Rare hereditary problems of galactose intolerance.
* Lactase enzyme deficiency or glucose galactose malabsorption
* Clinically significant abnormal level of serum creatinine
* Patients whose occupations make them unlikely to return to the clinic within 24h of treatment initiation
* Pregnancy or breast-feeding
* Investigational drug or immunomodulator treatment in the 30 days prior randomisation
* Prior enrollment in this study
* Participation in another therapeutic trial evaluating new drugs or which could interfere with the evolution of herpes labialis or the evaluation of the drug in the study within preceding 30 day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1727 (Actual)
Dates: Start 2007-05; Primary Completion 2008-11 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (53):
- United States (10):
  - Radiant Research, Inc.,, Scottsdale, Arizona
  - Radiant Research, Inc.,, Tucson, Arizona
  - Dermatology Private Practice, San Francisco, California
  - Front Range Clinical Research, Wheat Ridge, Colorado
  - St. Luke's Family Health,, Meridian, Idaho
  - Clinvest, a Division of Banyan Group, Inc.,, Springfield, Missouri
  - Rochester Clinical Research, Inc.,, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Center for Clinical Studies, Houston, Texas
  - Center for Clinical Studies, Ltd., LLP., Houston, Texas
- Australia (2):
  - Taylor Square Private Clinic, Sydney
  - Central Brunswick Medical Centre, Sydney
- Czechia (5):
  - General Teaching Hospital, Dep. Of Dermatology, Opava
  - U zastavky 16, Opava
  - Central military hospital Dept. of Dermatology, Prague
  - University Hospital Bulovka 3rd Clinic of Inf. Diseases, Prague
  - University Hospital Bulovka Dept. of Dermatology, Prague
- France (11):
  - Hôpital St Jacques Service de Dermatologie, Besançon
  - Private Practice, Martigues
  - Hopital Fournier, Service de dermatologie, Nancy
  - Private Practice, Nice
  - Hôpital L'Archet 2, Service de Dermatologie, Nice
  - Private Practice, Paris
  - Hôpital Tenon, Dermatology department, Paris
  - Hôpital Saint Louis Paris, Service de Dermatologie 1, Paris
  - Service de Stomatologie et chirurgie Maxilo-Faciale.Hôpital de la pitié Salpétrière, Paris
  - Hôpital Nord, Service de dermatologie, Saint-Etienne
  - Hôpital TROUSSEAU, Tours
- Germany (10):
  - Praxis Dres. Dörzapf und Partner, Augsburg
  - Charité Universitätsmedizin Berlin Klinik für Dermatologie, Venerologie und Allergologie, Berlin
  - Praxis, Berlin
  - Polikum Friedenau, Berlin
  - Gemeinschaftspraxis, Berlin
  - Laserclinic Drs. Steinert, Biberach
  - Klinik und Poliklinik für Dermatologie des Universitätsklinikums Bonn, Bonn
  - Praxis, Frankfurt
  - Raiffeisenstr. 15b, Oberkirch
  - Ludwig-Erhard-Platz 9-11, Rodgau-Dudenhofen
- Poland (10):
  - Katedra i Klinika Dermatologii Collegium Medicum, Bydgoszcz
  - Centrum Medyczne Diabet, Chrzanów
  - Naukowo-Badawczy i Naukowo-Dydaktyczny Ośrodek Dermatologii Estetycznej, Dermatochirurgii i Fotodermatologii, Gdynia
  - Niepubliczny Zaklad Opieki Zdrowotnej GCP Dobra Praktyka Lekarska, Grudziądz
  - NZOZ Atopia, Al. J., Krakow
  - Specjalistyczne Gabinety Lekarskie Dermed, Lodz
  - Niepubliczny Zakład Opieki Zdrowotnej Specjalistyczna Przychodnia Lekarska Medikard, Płock
  - Niepubliczny Zakład Opieki Zdrowotnej "Nasz Lekarz" Praktyka Grupowa Lekarzy Rodzinnych z Przychodnią Specjalistyczną, Torun
  - Gabinet Internistyczny, Warsaw
  - NZOZ Praktyka Lekarska Iga Gilas - Mirkiewicz, Wroclaw
- United Kingdom (5):
  - Cossington House Surgery, Canterbury
  - School of Dentistry, Cardiff University, Cardiff
  - Sidley Surgery, East Sussex
  - Sea Road Surgery, East Sussex
  - Saltash Health Centre, Saltash

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened beginning March 2007 and the last patient was treated in October 2008. The study was conducted at 47 sites in Australia, the Czech Republic, France, Germany, Poland, the United Kingdom and the United States.
Pre-assignment Details: Per protocol, a total of 1950 patients were to be randomized. Following randomization, patients were not to start treatment until a new labial herpes episode occurred. Thus, of those randomized, only 780 patients were planned to be treated (390 patients per treatment group) and 1170 patients were to be randomized, but not treated.
Groups:
- Acyclovir Lauriad Group: Acyclovir Lauriad 50mg muco-adhesive tablet
- Placebo Group: muco-adhesive buccal tablet with placebo
Period: Overall Study
Arm/Group | Acyclovir Lauriad Group | Placebo Group
Started | 378 (The number of participants started is defined as those that were randomized and received treatment.) | 397 (The number of participants started is defined as those that were randomized and received treatment.)
Completed | 361 | 384
Not Completed | 17 | 13

BASELINE CHARACTERISTICS:
Groups:
- Acyclovir Lauriad Group: Acyclovir Lauriad 50mg muco-adhesive tablet/Intent-to-Treat population
- Placebo Group: muco-adhesive buccal tablet with placebo/Intent-to-Treat population
- Total: Total of all reporting groups
Arm/Group | Acyclovir Lauriad Group | Placebo Group | Total
Number analyzed (Participants) | 376 | 395 | 771
Age Continuous [Mean (Standard Deviation); unit: years] — Data are provided for the Intent-to-Treat population.
  years | 40 (12.97) | 41.9 (13.33) | 41.0 (13.18)
Sex: Female, Male [Count of Participants; unit: Participants] — Data are provided for the Intent-to-Treat population.
  Participants
    Female | 258 | 271 | 529
    Male | 118 | 124 | 242
Region of Enrollment [Number; unit: participants] — Data are provided for the Intent-to-Treat population.
  participants
    United States | 71 | 72 | 143
    France | 41 | 49 | 90
    Czech Republic | 47 | 50 | 97
    Poland | 74 | 70 | 144
    Australia | 53 | 68 | 121
    Germany | 79 | 77 | 156
    United Kingdom | 11 | 9 | 20

OUTCOME MEASURES:

1. Secondary Outcome: Abortion of Primary Lesions
Description: Aborted lesions were defined as herpetic lesions preceded by prodromal symptoms that did not progress beyond the papule stage.
Time Frame: Assessed from the time of treatment initiation through Day 14
Population: This endpoint was analyzed using the Intent-to-Treat (ITT) population, which consisted of all randomized patients who received at least one dose of study medication and who had complete information recorded for the application time.
Measure: Number; unit: participants
Arm/Group | Acyclovir Lauriad Group | Placebo Group
Number analyzed (Participants) | 376 | 395
participants
  Aborted Lesions = Yes | 130 | 109
  Aborted Lesions = No | 242 | 279
  Aborted Lesions = Missing | 4 | 7
Statistical Analysis 1: Comparison: Acyclovir Lauriad Group vs Placebo Group; Test type: Superiority or Other; p = 0.0419, Chi-squared — p-value < 0.05 considered significant; Treatment difference = 0.0685, 95% CI 2-sided [0.0025 to 0.1339] — Treatment difference was the proportion of patients with aborted lesions in the acyclovir Lauriad group minus the proportion of patients with aborted lesions in the placebo group

2. Secondary Outcome: TTH of Non-primary Lesions (Aborted Lesions Excluded)
Description: TTH of non-primary lesions was defined as the time from treatment initiation to healing of all non-primary vesicular lesions. Non-primary lesions were those that developed in addition to and/or in 1 or more days after the primary vesicular lesion and that were located at least 1 cm from the primary lesion. Aborted lesions were not included in this parameter. TTH was to be assessed by the investigator.
Time Frame: Assessed from the time of treatment initiation through Day 14
Population: This endpoint was analyzed using a subgroup of patients in the ITT population with non-primary lesions.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Acyclovir Lauriad Group | Placebo Group
Number analyzed (Participants) | 39 | 62
Days | 7.00 [5.53 to 8.70] | 9.08 [7.46 to 11.00]
Statistical Analysis 1: Comparison: Acyclovir Lauriad Group vs Placebo Group; Test type: Superiority or Other; p = 0.0683, Log Rank — p-value < 0.05 considered significant

3. Secondary Outcome: Duration of Episode (DOE)
Description: For patients who experienced a vesicular lesion, DOE was defined as the time from treatment initiation to healing of primary and secondary vesicular lesions (loss of crust). For subjects whose primary and secondary lesions were not vesicular in nature, DOE was defied as the time from treatment initiation to return to normal skin or to cessation of symptoms, whichever came last.
Time Frame: Assessed from initiation of treatment to Day 14
Population: This endpoint was analyzed using the ITT population.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Acyclovir Lauriad Group | Placebo Group
Number analyzed (Participants) | 373 | 395
Days | 5.57 [5.03 to 6.01] | 6.38 [5.93 to 6.97]
Statistical Analysis 1: Comparison: Acyclovir Lauriad Group vs Placebo Group; Test type: Superiority or Other; p = 0.0033, Log Rank — p-value < 0.05 considered significant

4. Secondary Outcome: Time to Cessation of Symptoms
Description: Time to cessation of symptoms was defined as the time from treatment initiation to cessation of all symptoms: pain, burning, itching, tingling, tenderness and discomfort. It was to be assessed by the investigator.
Time Frame: Assessed from time of treatment initiation through Day 14
Population: This endpoint was analyzed using the ITT population.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Acyclovir Lauriad Group | Placebo Group
Number analyzed (Participants) | 373 | 393
Days | 3.57 [3.04 to 4.01] | 4.16 [3.75 to 4.89]
Statistical Analysis 1: Comparison: Acyclovir Lauriad Group vs Placebo Group; Test type: Superiority or Other; p = 0.0098, Log Rank — p-value < 0.05 considered significant

5. Secondary Outcome: TTH of Aborted Primary Lesions
Description: TTH of aborted primary lesions was defined as the time from treatment initiation to healing of the primary lesion (erythema or papule) or cessation of symptoms, whichever came last. It was to be assessed by the investigator.
Time Frame: Assessed from time of treatment initiation through Day 14
Population: This endpoint was analyzed using the subgroup of patients within the ITT population with aborted lesions.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Acyclovir Lauriad Group | Placebo Group
Number analyzed (Participants) | 108 | 85
Days | 2.57 [2.00 to 2.96] | 2.67 [2.10 to 3.04]
Statistical Analysis 1: Comparison: Acyclovir Lauriad Group vs Placebo Group; Test type: Superiority or Other; p = 0.8005, Log Rank — p-value < 0.05 considered significant

6. Primary Outcome: Time to Healing (TTH) of Vesicular Primary Lesion
Description: Healing was defined as the loss of crust (erythema may be present) as assessed by the investigator. TTH was the time from treatment initiation to healing as defined above and was assessed from the time of treatment initiation through Day 14. The primary vesicular lesion was the first developed lesion located on the lip and was not to have extended more than 1 cm outside the lip.
Time Frame: Assessed from time of treatment initiation through Day 14
Population: The modified Intent-to-Treat (mITT) population was the population used for analysis of this endpoint. The mITT population included all randomized patients who received at least one dose of study medication and who reached the vesicular stage (ie, episodes that progressed through macula, papule, vesicle, crust and healing).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Acyclovir Lauriad Group | Placebo Group
Number analyzed (Participants) | 242 | 279
Days | 7.00 (0.18) [6.75 to 7.31] | 7.32 (0.18) [6.97 to 7.92]
Statistical Analysis 1: Comparison: Acyclovir Lauriad Group vs Placebo Group; Test type: Superiority or Other; p = 0.015, Log Rank — p-value < 0.05 considered significant

7. Secondary Outcome: Time to Recurrence of Non-aborted Lesions During 9-month Follow-up
Description: Time to recurrence was the time from the healing of all lesions of the initial episode to the occurrence of new lesions.
Time Frame: From time of initial healing through the 9-month follow-up
Population: This endpoint was analyzed using the follow-up population, a subgroup of the ITT population who continued to the 9 month follow-up and had at least 1 diary assessment during that period. The follow-up population was defined as patients whose lesions were healed at the end of Day 14 and had no recurrence within 15 days of healing of all lesions.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Acyclovir Lauriad Group | Placebo Group
Number analyzed (Participants) | 232 | 246
Days | 205.0 (19.4) [163.0 to 287.0] | 165.0 (9.3) [136.0 to 203.0]
Statistical Analysis 1: Comparison: Acyclovir Lauriad Group vs Placebo Group; Test type: Superiority or Other; p = 0.0412, Log Rank — p-value < 0.05 considered significant

8. Secondary Outcome: Patient Incidence of Recurrence of Non-aborted Lesions During 9-month Follow-up
Description: Recurrence was the occurrence of new lesions and was evaluated in a subgroup of patients who agreed to record recurrences during the 9-month follow-up period.
Time Frame: From time of initial healing through the 9-month follow-up
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Acyclovir Lauriad Group | Placebo Group
Number analyzed (Participants) | 267 | 270
participants
  Recurrence during 9-month follow-up = yes | 149 | 181
  Recurrence during 9-month follow-up = no | 83 | 65
  Recurrence during 9-month follow-up = missing | 35 | 24
Statistical Analysis 1: Comparison: Acyclovir Lauriad Group vs Placebo Group; Test type: Superiority or Other; p = 0.0271, Chi-squared — p-value < 0.05 considered significant

9. Secondary Outcome: Symptom Intensity (Visual Analogue Scale [VAS])
Description: Patients were asked to place a tick mark on a 10 centimeter VAS indicating their symptom intensity. Scale ratings ranged from a minimum of 0 (none at all) to a maximum of 10 (worst possible). The location of the tick mark from "0" was measured in millimeters (0 - 100) and recorded.
Time Frame: Assessed on Days 1, 3, 5, 7 and 14 (or within 24 hours of healing)
Population: This endpoint was analyzed using the safety population, which consisted of all randomized patients who took at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale (0 - 100)
Arm/Group | Acyclovir Lauriad Group | Placebo Group
Number analyzed (Participants) | 378 | 397
units on a scale (0 - 100)
  Day 1 | 30.5 (22.37) | 31.1 (22.07)
  Day 3 | 21.2 (22.88) | 22.9 (22.60)
  Day 5 | 12.7 (17.60) | 17.3 (20.70)
  Day 7 | 8.2 (13.63) | 10.7 (18.48)
  Day 14 (or within 24 hours of healing) | 1.0 (5.14) | 0.9 (3.61)
Statistical Analysis 1: Comparison: Acyclovir Lauriad Group vs Placebo Group; Analysis conducted between treatment groups at Day 1 timepoint; Test type: Superiority or Other; p = 0.5695, Wilcoxon (Mann-Whitney) — p-value < 0.05 considered significant
Statistical Analysis 2: Comparison: Acyclovir Lauriad Group vs Placebo Group; Analysis conducted between treatment groups at Day 3 timepoint; Test type: Superiority or Other; p = 0.1824, Wilcoxon (Mann-Whitney) — p-value < 0.05 considered significant
Statistical Analysis 3: Comparison: Acyclovir Lauriad Group vs Placebo Group; Analysis conducted between treatment groups at the Day 5 timepoint; Test type: Superiority or Other; p = 0.0078, Wilcoxon (Mann-Whitney) — p-value < 0.05 considered significant
Statistical Analysis 4: Comparison: Acyclovir Lauriad Group vs Placebo Group; Analysis conducted between treatment groups at the Day 7 timepoint; Test type: Superiority or Other; p = 0.3303, Wilcoxon (Mann-Whitney) — p-value < 0.05 considered significant
Statistical Analysis 5: Comparison: Acyclovir Lauriad Group vs Placebo Group; Analysis conducted between treatment groups at the Day 14 timepoint; Test type: Superiority or Other; p = 0.6045, Wilcoxon (Mann-Whitney) — p-value < 0.05 considered significant

10. Secondary Outcome: Patient Satisfaction With Treatment
Description: At the end of study (Day 14 [or within 24 hours of healing]), patients were asked whether they were satisfied with treatment (yes/no).
Time Frame: Assessed on Day 14 (or within 24 hours of healing)
Population: This endpoint was analyzed using the ITT population.
Measure: Number; unit: participants
Arm/Group | Acyclovir Lauriad Group | Placebo Group
Number analyzed (Participants) | 376 | 395
participants
  Satisfied with treatment = yes | 297 | 275
  Satisfied with treatment = no | 66 | 105
  Missing | 13 | 15
Statistical Analysis 1: Comparison: Acyclovir Lauriad Group vs Placebo Group; Test type: Superiority or Other; p = 0.0022, Chi-squared — p-value < 0.05 considered significant

11. Secondary Outcome: Patient Assessment of Efficacy of the Treatment
Description: At the end of study (Day 14 [ or within 24 hours of healing]), patients were asked to rate efficacy of treatment using a 4-point scale (inactive, mildly active, moderately active, or very active).
Time Frame: Assessed on Day 14 (or within 24 hours of healing)
Population: This endpoint was analyzed using the ITT population.
Measure: Number; unit: participants
Arm/Group | Acyclovir Lauriad Group | Placebo Group
Number analyzed (Participants) | 376 | 395
participants
  Inactive | 50 | 79
  Midly active | 49 | 44
  Moderately active | 100 | 104
  Very active | 154 | 146
  Missing | 23 | 22

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during the 14 day treatment period.
Description: The safety population included all randomized patients who took at least 1 dose of study drug, including 378 patients in the acyclovir Lauriad group and 397 patients in the placebo group.
Arm/Group | Acyclovir Lauriad Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/378 | 1/397
Other Adverse Events (participants affected / at risk) | 20/378 | 22/397
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acyclovir Lauriad Group (N=378) | Placebo Group (N=397)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acyclovir Lauriad Group (N=378) | Placebo Group (N=397)
headache (Nervous system disorders) | 12 (12) | 12 (12)
Nasopharyngitis (Infections and infestations) | 4 (4) | 3 (3)
Application Site Pain (General disorders) | 4 (4) | 4 (4)
nausea (Gastrointestinal disorders) | 1 (1) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less